CLINICAL TRIAL: NCT00068081
Title: A Randomized, Double-Blind, Controlled Study of NGX-4010 for the Treatment of Postherpetic Neuralgia
Brief Title: Controlled Study of NGX-4010 for the Treatment of Postherpetic Neuralgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NeurogesX (Industry)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: C110
Record Dates: First submitted 2003-09-05; First posted 2003-09-09 (Estimated); Last update posted 2008-03-06 (Estimated); Status verified 2007-09

CONDITIONS: Herpes Zoster; Neuralgia; Pain; Peripheral Nervous System Diseases
Keywords: Dermal assessment; Pain measurement; Diary; Analgesics/*therapeutic use; Capsaicin/*administration & dosage/adverse effects; Herpes zoster/*complication/drug therapy; Neuralgia/*drug therapy/etiology; Pain; Peripheral nervous system diseases/*complications
MeSH Terms: conditions — Herpes Zoster; Neuralgia; Pain; Peripheral Nervous System Diseases

INTERVENTIONS:
Drug: Capsaicin Dermal Patch

SUMMARY:
The purpose of the study is to assess the efficacy, safety and tolerability of NGX 4010 applied for 60 minutes for the treatment of PHN.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Be in good health.
* Diagnosis of postherpetic neuralgia (PHN) made by the primary treating physician or Investigator, and at least 3 months post-vesicle crusting.
* Screening Pain Sum Score of 12 to 36.
* Intact, unbroken skin over the painful area(s) to be treated.
* If taking chronic pain medications, be on a stable (not PRN) regimen for at least 21 days prior to Treatment Visit (Day 0) and willing to maintain medications at same stable dose(s) and schedule throughout the study.
* Female subjects with child-bearing potential must have a negative serum beta hCG pregnancy test, to be performed at the Screening Visit.
* All subjects must be willing to use effective methods of birth control and/or refrain from participating in a conception process during the study and for 30 days following experimental drug exposure.
* Be willing and able to comply with protocol requirements for the duration of study participation. (Such requirements include, but are not limited to: completing a daily pain diary, attending all study visits, and refraining from elective surgery and extensive travel during study participation.)

Exclusion Criteria:

* Concomitant opioid medication, unless orally or transdermally administered and not exceeding a total daily dose of morphine 60 mg/day, or equivalent. Parenteral opioid use is excluded, regardless of dose.
* Unavailability of an effective rescue medication strategy for the subject, such as unwillingness to use opioid analgesics during treatment, or high tolerance to opioids precluding the ability to relieve treatment-associated discomfort with Roxicodone®, as judged by the Investigator.
* Active substance abuse or history of chronic substance abuse within the past year, or prior chronic substance abuse judged likely to recur during the study period by the investigator.
* Recent use (within 21 days preceding the Treatment Visit [Day 0]) of any topically applied pain medication, such as non-steroidal anti-inflammatory drugs, menthol, methyl salicylate, local anesthetics (including Lidoderm®), steroids or capsaicin products on the painful areas.
* Current use of any investigational agent, or Class 1 anti-arrhythmic drugs (such as tocainide and mexiletine).
* Significant pain of an etiology other than PHN, for example, compression-related neuropathies (e.g., spinal stenosis) or fibromyalgia or arthritis. Subjects must not have significant ongoing pain from other cause(s) that may interfere with judging PHN-related pain.
* Painful PHN areas located only on the face, above the hairline of the scalp, and/or in proximity to mucous membranes. (Investigational treatment with NGX-4010 is not allowed in these areas.)
* Any implanted medical device (spinal cord stimulator, intrathecal pump or peripheral nerve stimulator) for the treatment of neuropathic pain.
* Hypersensitivity to capsaicin (i.e., chili peppers or Over-the-Counter (OTC) capsaicin products), local anesthetics, Roxicodone® or adhesives.
* Significant ongoing or untreated abnormalities in cardiac, renal, hepatic, or pulmonary function that may interfere either with the ability to complete the study or the evaluation of adverse events.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - NeurogesX Investigational Site, Mesa, Arizona
  - NeurogesX Investigational Site, Peoria, Arizona
  - NeurogesX Investigational Site, Phoenix, Arizona
  - NeurogesX Investigational Site, Duarte, California
  - NeurogesX Investigational Site, Santa Rosa, California
  - NeurogesX Investigational Site, Boynton Beach, Florida
  - NeurogesX Investigational Site, Bradenton, Florida
  - NeurogesX Investigational Site, Fort Myers, Florida
  - NeurogesX Investigational Site, Naples, Florida
  - NeurogesX Investigational Site, Tampa, Florida
  - NeurogesX Investigational Site, Atlanta, Georgia
  - NeurogesX Investigational Site, Marietta, Georgia
  - NeurogesX Investigational Site, Brighton, Massachusetts
  - NeurogesX Investigational Site, St Louis, Missouri
  - NeurogesX Investigational Site, Winston-Salem, North Carolina
  - NeurogesX Investigational Site, Dallas, Texas
  - NeurogesX Investigational Site, San Antonio, Texas
  - NeurogesX Investigational Site, Salt Lake City, Utah

REFERENCES:
- [Derived] Webster LR, Tark M, Rauck R, Tobias JK, Vanhove GF. Effect of duration of postherpetic neuralgia on efficacy analyses in a multicenter, randomized, controlled study of NGX-4010, an 8% capsaicin patch evaluated for the treatment of postherpetic neuralgia. BMC Neurol. 2010 Oct 11;10:92. doi: 10.1186/1471-2377-10-92. PMID 20937130